CLINICAL TRIAL: NCT06838091
Title: Effect of Low-Flow Anesthesia in Single Lung Ventilation on Postoperative Respiratory Complications
Acronym: Low-Flow Anest
Status: Completed | Type: Observational
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Cansu KILINC BERKTAS, Specialist Doctor, Başakşehir Çam & Sakura City Hospital
Other Study IDs: 243
Record Dates: First submitted 2025-02-12; First posted 2025-02-20 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-02

CONDITIONS: Thoracic Surgery; Low-flow Anesthesia
Keywords: Low-flow anesthesia; thoracic surgery
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (4):
- group 1: 0.5 lt/min
  Interventions: Other: Observational
- group 2: 0.5-1 lt/min
  Interventions: Other: Observational
- group 3: 1-2 lt/min
  Interventions: Other: Observational
- group 4: > 2lt/min
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — During anesthesia administration:
  T0, T1, T2, T3, T4 represent the following periods:
  T0: Double lumen ventilation in the supine position immediately after intubation T1: Double lumen ventilation in the lateral position T2: Single lumen ventilation in the lateral position (with the chest wall closed) T3: Single lumen ventilation in the lateral position (with the chest wall open) T4: Just before extubation
  1. Airway pressure (P plateau, Ppeak) values from the anesthesia device data,
  2. BIS (from routine BIS monitoring)
  3. Temperature (Routinely from pharyngeal temperature probe),
  4. Oxygen saturation (Routinely from the patient monitor)
  5. End-tidal CO₂,
  6. Inspiratory O₂ concentration,
  7. Inspiratory CO2 concentration,
  8. Inspiratory and expiratory desflurane/sevoflurane concentrations,
  9. Tidal volume,
  10. MAC, routinely from anesthesia device data
  11. Blood Gas Analysis (COHgb, Ph, PO 2 , PCO 2 , SaO 2, HCO 3 , Base deficit, glucose, lactate)

SUMMARY:
Mechanical ventilation in thoracic surgery patients is often complicated because patients are usually in the lateral decubitus position and the operated lung is intermittently deflated to facilitate surgical exposure . Single-lung ventilation during thoracic surgery is prone to volutrauma, barotrauma, atelectrauma, and oxygen toxicity, which are important aspects of ventilator-associated lung injury (VILI) . In studies conducted on operated patients, the use of lung-protective ventilation, including low tidal volume (6-8 ml/kg), respiratory rate, driving pressure (DP), and positive end-expiratory pressure (PEEP) application, has been recommended in the perioperative period to reduce postoperative pulmonary complications. Optimum oxygenation should be provided to patients during the intraoperative period, avoiding the harmful effects of hypoxia and hyperoxia. This situation becomes even more important in single-lung ventilation. Fresh gas flow in anesthesia systems can be done with traditional high-flow, normal-flow, or low-flow strategies according to the clinician's preference. The interest in the anesthesia method with low fresh gas flow has increased all over the world and in our country. The development of the technology of the anesthesia devices used, the increase in knowledge about the content of inhaled gases, and the availability of monitors that continuously and thoroughly analyze the anesthetic gas composition have facilitated the use of low-flow anesthesia safely.

When the literature is evaluated, it is defined as 4 lt/min and above as very high flow, 2-4 lt/min as high flow, 1-2 lt/min as medium flow, 0.5-1 lt/min as low flow, 0.25-0.5 lt/min as minimal flow, and <0.25 lt/min as metabolic flow . High flow has now been abandoned due to both cost and environmental pollution.

Low-flow anesthesia creates a breath air closer to physiological conditions during anesthesia by heating and humidifying the inhaled gases. In addition, it provides a cost advantage by reducing inhalation agent consumption and reduces atmospheric pollution . It is suggested that the use of both fresh gas flow rates does not pose a safety risk for patients, and in fact, the use of low-flow anesthesia methods should be made more widespread with the advantages it provides. Low-flow anesthesia is a method applied during general anesthesia using a rebreathing anesthesia system, where the rebreathed fresh oxygen flow rate is at least 50%, metabolic requirements are fully met and sufficient volatile matter can be administered. In our clinic, the fresh gas flow rate during general anesthesia is routinely used at a value between 0.5 lt/min-3 lt/min, depending on the clinician's preference. In our clinic, low-flow anesthesia methods (with varying flows) are routinely applied in addition to normal flow methods in many surgical practices.

Although low-flow anesthesia techniques are used in many surgical practices, the literature is limited in surgeries where single-lung ventilation is performed. The purpose of this study is to determine the anesthetic flows used in amounts ranging from 0.5 lt/min-3 lt/min in thoracic surgeries where single-lung ventilation is performed; to evaluate the effects on perioperative hemodynamic and respiratory parameters and respiratory complications. The secondary aim of the study is to show the consumption of inhalation agent and soda lime.

DETAILED DESCRIPTION:
Mechanical ventilation in thoracic surgery patients is often complicated because patients are usually in the lateral decubitus position and the operated lung is intermittently deflated to facilitate surgical exposure. Single-lung ventilation during thoracic surgery is prone to volutrauma, barotrauma, atelectrauma, and oxygen toxicity, which are important aspects of ventilator-associated lung injury (VILI). In studies conducted on operated patients, the use of lung-protective ventilation, including low tidal volume (6-8 ml/kg), respiratory rate, driving pressure (DP), and positive end-expiratory pressure (PEEP) application, has been recommended in the perioperative period to reduce postoperative pulmonary complications. Optimum oxygenation should be provided to patients during the intraoperative period, avoiding the harmful effects of hypoxia and hyperoxia. This situation becomes even more important in single-lung ventilation. Fresh gas flow in anesthesia systems can be done with traditional high-flow, normal-flow, or low-flow strategies according to the clinician's preference. The interest in the anesthesia method with low fresh gas flow has increased all over the world and in our country. The development of the technology of the anesthesia devices used, the increase in knowledge about the content of inhaled gases, and the availability of monitors that continuously and thoroughly analyze the anesthetic gas composition have facilitated the use of low-flow anesthesia safely.

When the literature is evaluated, it is defined as 4 lt/min and above as very high flow, 2-4 lt/min as high flow, 1-2 lt/min as medium flow, 0.5-1 lt/min as low flow, 0.25-0.5 lt/min as minimal flow, and <0.25 lt/min as metabolic flow. High flow has now been abandoned due to both cost and environmental pollution.

Low-flow anesthesia creates a breath air closer to physiological conditions during anesthesia by heating and humidifying the inhaled gases. In addition, it provides a cost advantage by reducing inhalation agent consumption and reduces atmospheric pollution. It is suggested that the use of both fresh gas flow rates does not pose a safety risk for patients, and in fact, the use of low-flow anesthesia methods should be made more widespread with the advantages it provides. Low-flow anesthesia is a method applied during general anesthesia using a rebreathing anesthesia system, where the rebreathed fresh oxygen flow rate is at least 50%, metabolic requirements are fully met and sufficient volatile matter can be administered. In our clinic, the fresh gas flow rate during general anesthesia is routinely used at a value between 0.5 lt/min-3 lt/min, depending on the clinician's preference. In our clinic, low-flow anesthesia methods (with varying flows) are routinely applied in addition to normal flow methods in many surgical practices.

Although low-flow anesthesia techniques are used in many surgical practices, the literature is limited in surgeries where single-lung ventilation is performed. The purpose of this study is to determine the anesthetic flows used in amounts ranging from 0.5 lt/min-3 lt/min in thoracic surgeries where single-lung ventilation is performed; to evaluate the effects on perioperative hemodynamic and respiratory parameters and respiratory complications. The secondary aim of the study is to show the consumption of inhalation agent and soda lime.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo thoracic surgery with single lung ventilation
* ASA I-II-III class
* 18-75 years old
* Those who have received informed consent form approval

Exclusion Criteria:

* COPD and asthma diagnosis
* History of previous thoracic surgery
* Body mass index (BMI) >35
* Development of hemodynamic instability or desaturation during surgery (SpO2<92)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who will undergo thoracic surgery with single lung ventilation, ASA I-II-III class, 18-75 years old
Sampling Method: Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-02 (Actual)

PRIMARY OUTCOMES:
The effects of anesthetic flows varying | 01.03.2025- 01.06.2025
  Primary outcome is the effects of anesthetic flows varying between 0.5 lt/min-3 lt/min on perioperative hemodynamic and respiratory parameters and respiratory complications in thoracic surgeries with single lung ventilation.

CONTACTS AND LOCATIONS:
Locations (1):
- Başakşehir Çam Ve Sakura Şehir Hastanesi, Istanbul, İ̇stanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Because it is not completed